CLINICAL TRIAL: NCT05967988
Title: AtmosphEric pRojection for paIn and Anxiety reLated to Minor Medical Procedures in the Emergency Department: a Monocentric, Parallel, Randomized, Controlled Study
Brief Title: Atmospheric Projection in the Emergency Department
Acronym: AERIAL-MED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of resources
Sponsor: University of Lausanne Hospitals (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Principal Investigator, Olivier Hugli, Head of Emergency Department, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER-VD 2023-00867
Record Dates: First submitted 2023-06-28; First posted 2023-08-01 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pain, Acute; Anxiety Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient will assess the outcome him/herself. The statistician will also be blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atmospheric 3D video projection (Experimental): Patients in the interventional arm will watch an immersive atmospheric video projection on the walls of their examination room.
  Interventions: Device: Immersive atmospheric projection
- Atmospheric 3D color projection (Sham Comparator): Patients in the interventional arm will look at a neutral color of their choice projected on the walls of their examination room.
  Interventions: Device: Minimal atmospheric projection

INTERVENTIONS:
Device: Immersive atmospheric projection — Projection of computer-generated videos or videos of real moving landscapes on the walls of the examination room
  Arms: Atmospheric 3D video projection
Device: Minimal atmospheric projection — Projection of a colors on the walls on the walls of the examination room
  Arms: Atmospheric 3D color projection

SUMMARY:
The goal of this clinical trial is to learn about the reduction of pain and anxiety during a minor procedure in the emergency department on adult patients through the visualisation of atmospheric projection as a distraction mean. The main question it aims to answer is :

Can the atmospheric projection of a video reduce pain and anxiety in adult patients receiving painful procedures in the emergency department ?

Participants will look at an atmospheric projection (projection of a media on the walls and roof around the patient) while receiving their planned care procedures. Researchers will compare an active group watching a video with a control group watching a simple colored light to see if the visualisation of an atmospheric projected video reduces pain and anxiety more than the visualisation of a colored light does.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 ;
* Patient requiring one of the following treatment procedures : suturing, plaster cast placement and/or repositioning, fracture or dislocation reduction, ascites puncture, pleural puncture, lumbar puncture.

Exclusion Criteria:

* Patient clinically unstable;
* Patient incapable of discernment or consent ;
* Altered mental status (cognitive disorders, mental retardation, acute state of confusion, acute psychosis);
* Alcoholic patient with University of California, San Diego Brief Assessment of Capacity to Consent (UBACC) score of 10/10 ;
* Patient hard of hearing ;
* Patient with visual impairments preventing him/her from perceiving his/her environment ;
* Patient unable to understand the use of visual analog scales (VAS);
* Impaired sensitivity of the part of the body where the medical intervention is to take place;
* Planned use of analgesia/sedation with a dissociative agent (midazolam, ketamine, propofol);
* Incarcerated patient ;
* Patient transferred from another hospital ;
* Patient having already participated in this study during a previous consultation in the emergency department of the Centre Hospitalier Universitaire Vaudois.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Procedural Pain | Just after the procedure
  Maximal pain intensity experienced by the patient during the medical procedure, assessed using a Visual Analogic Scale from 0mm to 100mm anchored with "No pain/Worst pain imaginable"
Procedural Anxiety | Just after the procedure
  Maximal anxiety intensity felt by the patient during the medical procedure, assessed using a Visual Analogic Scale from 0mm to 100mm anchored with "Not at all anxious/Extremely anxious."

SECONDARY OUTCOMES:
Telepresence | Just after the procedure
  Telepresence will be assessed by the Igroupe Presence Questionnaire composed of 14 statements grouped into 4 categories: (1) spatial presence (the sense of being physically present in the virtual environment), (2) involvement (attention devoted to the virtual environment and experienced involvement), (3) experienced realism (the subjective experience of realism in the virtual environment), and (4) the general sense of being in the virtual environment. Each question is rated on a 7-point scale (0 to 6), with greater scores indicating a greater sense of presence in the projected environment
Dissociation | Just after the procedure
  Dissociation of the patients represents the mental separation of the patient from their environment, assessed using a Visual Analogic Scale from 0mm to 100mm, anchored with "most present in the clinical environment / the most immersed in the projected environment "
Appreciation of the atmospheric projection | Just after the procedure
  Appreciation of the atmospheric projection by the patient, using a Visual Analogic Scale from 0mm to 100mm, anchored with "least appreciative/most appreciative)
Patient's comfort | Just after the procedure
  Patient's comfort during the atmospheric projection, assessed using a Visual Analogic Scale from 0mm to 100mm, anchored with "least comfortable /most comfortable"
Procedural support | After the procedure
  Procedural support provided by the projection during the medical procedure according to the physician in charge of the procedure, assessed using a 3-level Likert scale (yes-neutral-no)
Procedural disturbance | Just after the procedure
  Procedural disturbance for physicians caused by the atmospheric projection interfering with the medical procedure, assessed using a 3-level Likert scale (yes-neutral-no)
Cybercinetosis | Just after the procedure
  Cybercinetosis is a symptom similar to motion sickness that occurs with exposure to a virtual environment, will be assessed using a 3-level Likert scale (light-moderate-severe)
Pain catastrophizing | Just before the procedure
  Pain catastrophizing will be assessed using the French version of the Situational Catastrophizing Questionnaire, a 6-question adaptation of the Pain Catastrophizing Scale

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hugli, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No